CLINICAL TRIAL: NCT00496626
Title: An Immunogenicity and Safety Study of Quadrivalent HPV (Types 6, 11, 16, 18) Virus-Like Particle (VLP) Vaccine in Chinese Female Subjects Aged 9 to 45 Years and Male Subjects Aged 9 to 15 Years
Brief Title: An Immunogenicity and Safety Study of Gardasil® in Chinese Subjects (V501-030)(COMPLETED)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V501-030; 2007_021; NCT00926822 (obsolete NCT alias)
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Results first posted 2010-07-09 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-03

CONDITIONS: Papillomavirus Infections
Keywords: HPV infections
MeSH Terms: conditions — Papillomavirus Infections | interventions — Papillomavirus Vaccines; Vaccines, Synthetic; Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): V501 (Gardasil®)
  Interventions: Biological: Quadrivalent Human Papillomavirus (HPV, Types 6, 11, 16, 18) Recombinant Vaccine (Gardasil®)
- 2 (Placebo Comparator): Placebo
  Interventions: Biological: Comparator: Placebo

INTERVENTIONS:
Biological: Quadrivalent Human Papillomavirus (HPV, Types 6, 11, 16, 18) Recombinant Vaccine (Gardasil®) — Human Papillomavirus (Type 6, 11, 16, 18) Recombinant Vaccine (Gardasil®), 0.5mL, 3 Dose of intramuscular injection at Day 1, Month 2 and Month 6
  Other Names: V501; Gardasil®
  Arms: 1
Biological: Comparator: Placebo — aluminum-contained, 0.5mL, 3 Dose of intramuscular injection at Day 1, Month 2 and Month 6
  Arms: 2

SUMMARY:
This is a China registration study. A randomized, double-blind, placebo-controlled immunogenicity and safety study in Chinese female participants aged 9 to 45 years and male participants aged 9 to 15 years. Approximately 600 participants will be randomized in a 1:1 ratio to receive either vaccine or aluminum-containing placebo. Each participant received one injection at each visit at Day 1, Month 2, and Month 6. Vaccine or placebo was given as a 0.5-mL intramuscular injection. Serum will be collected from all participants to evaluate immune response against anti-Human Papillomavirus (HPV) 6/11/16/18 with Luminex Assay. At Month 2, Month 6, Month 7, subjects will be evaluated for any new medical condition or health concerns and Serious Adverse Experiences throughout the study. The primary objective is to evaluate the vaccine-induced serum anti-HPV 6, 11, 16 and 18 antibody titers following 3-dose regimen of Gardasil® compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female participants aged 9-45 years old and male participants aged 9-15 years old
* Participants agrees to provide study personnel with a primary telephone number as well as an alternate telephone number for follow-up purposes
* Not pregnant now (as demonstrated by a negative urine beta-Human Chorionic Gonadotropin (beta-HCG) test) for post-pubertal female participants

Ages: 9 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 600 (Actual)
Dates: Start 2008-07-20 (Actual); Primary Completion 2009-02-28 (Actual); Study Completion 2009-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Li R, Li Y, Radley D, Liu Y, Huang T, Sings HL, Zhang L, Wang W, Zhong X, Saah AJ. Safety and immunogenicity of a vaccine targeting human papillomavirus types 6, 11, 16 and 18: a randomized, double-blind, placebo-controlled trial in Chinese males and females. Vaccine. 2012 Jun 13;30(28):4284-91. doi: 10.1016/j.vaccine.2012.02.079. Epub 2012 Mar 18. PMID 22433961
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263

RESULTS

PARTICIPANT FLOW:
Groups:
- Vaccine (Gardasil®) Group: Human Papillomavirus (HPV) (Type 6, 11, 16, 18) Recombinant Vaccine (Gardasil®), 0.5mL, 3 Dose of intramuscular injection at Day 1, Month 2 and Month 6
- Placebo Group: Placebo aluminum-containing, 0.5mL, 3 Dose of intramuscular injection at Day 1, Month 2 and Month 6
Period: Overall Study
Arm/Group | Vaccine (Gardasil®) Group | Placebo Group
Started | 302 | 298
Completed | 296 | 292
Not Completed | 6 | 6
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 5 | 4
Not completed — Relocated | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vaccine (Gardasil®) Group | Placebo Group | Total
Number analyzed (Participants) | 302 | 298 | 600
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.5 (10.9) | 24.8 (11.0) | 24.6 (10.9)
Age, Customized [Number; unit: Participants]
  9-15 Years of Age | 101 | 99 | 200
  16-26 Years of Age | 76 | 74 | 150
  27-34 Years of Age | 63 | 62 | 125
  35-45 Years of Age | 62 | 63 | 125
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 251 | 249 | 500
  Male | 51 | 49 | 100
Body Temperature [Mean (Standard Deviation); unit: Degrees Celsius] | 36.5 (0.31) | 36.5 (0.31) | 36.5 (0.31)
Pulse [Mean (Standard Deviation); unit: Beats per minute (BPM)] | 74.4 (11.9) | 74.6 (11.2) | 74.5 (11.2)

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titer (GMT) of Anti-HPV 6, 11, 16 , 18 at Day 1 and Month 7 (1 Month After Completion of Administration of a 6-month 3-dose Regimen of Vaccines)
Description: Measured GMT of anti-HPV 6, 11, 16 and 18 at Day 1 and Month 7 (1 month after completion of administration of a 6-month 3-dose regimen of vaccines). GMT at Day 1 was used to define per-protocol population. Antibody titers were tested with Luminex array.
  The numeric values for the Day 1 (Vaccine and Placebo groups) and the Month 7 (Placebo groups) are the threshold of detection for the Luminex array assays. The reported values are all below the lower limit of qualification, ((less than) <7, <8, <11, <10 respectively)
Time Frame: Collect blood sample for anti-HPV 6, 11, 16, 18 titers testing at Day 1 prior to vaccination, and Month 7
Population: Per-protocol population, defined as all participants who received all 3 dose vaccinations within acceptable day ranges, had at least 1 valid serology result after the third injection, and adhered to protocol guidelines. To be included in the immunogenicity analysis for given HPV type, participants must be seronegative to that HPV type at baseline.
Measure: Geometric Mean (95% Confidence Interval); unit: mMU/mL
Groups:
- Vaccine (Gardasil®) Group (Day 1); Vaccine (Gardasil®) Group (Month 7): Human Papillomavirus (HPV) (Type 6, 11, 16, 18) Recombinant Vaccine (Gardasil®), 0.5mL, 3 Dose of intramuscular injection at Day 1, Month 2 and Month 6
- Placebo Group (Day 1); Placebo Group (Month 7): Placebo aluminum-containing, 0.5mL, 3 Dose of intramuscular injection at Day 1, Month 2 and Month 6
Arm/Group | Vaccine (Gardasil®) Group (Day 1) | Placebo Group (Day 1) | Vaccine (Gardasil®) Group (Month 7) | Placebo Group (Month 7)
Number analyzed (Participants) | 302 | 298 | 302 | 298
mMU/mL
  anti-HPV 6 | 7 [7 to 7] | 7 [7 to 7] | 426.0 [369.5 to 491.0] | 7 [7 to 7]
  anti-HPV 11 | 8 [8 to 8] | 8 [8 to 8] | 665.0 [589.4 to 750.3] | 8 [8 to 8]
  anti-HPV 16 | 11 [11 to 11] | 11 [11 to 11] | 2336.9 [2023.1 to 2699.3] | 11 [11 to 11]
  anti-HPV 18 | 10 [10 to 10] | 10 [10 to 10] | 535.6 [461.8 to 621.2] | 10 [10 to 10]
Statistical Analysis 1: Comparison: Vaccine (Gardasil®) Group (Month 7) vs Placebo Group (Month 7); An Analysis of Covariance (ANCOVA) model was used for each HPV type, based on the pooled data from all age groups and genders. The natural-log-transformed titer was the response variable, and vaccination group, gender and age group were covariates. The null hypothesis was that the GMT ratio (Gardasil/Placebo) was equal to 1; Test type: Superiority or Other; p <= 0.05, ANCOVA — The ANCOVA models showed the lower bounds of two-sided 95% CI on the GMT ratio [GARDASIL™/placebo] were greater than 1 for each HPV type, so the null hypothesis was rejected. The CI reported is for HPV18, the type with the smallest CI lower bound; GMT ratio = 101.6, 95% CI 2-sided [88.1 to 117.2] — Superiority of GARDASIL™ to placebo was claimed if, for each of the four HPV types, the lower bound of the two-sided 95% CI on the GMT ratio [GARDASIL™/placebo] being >1, or equivalently, the two-sided p-value <0.05

2. Secondary Outcome: Number of Participants Who Were Seronegative at Baseline and Developed Seropositive at Month 7
Description: Anti-HPV 6, 11, 16, 18 Seroconversion Rate, i.e., the Number of participants who were seronegative at baseline and developed seropositive at Month 7. Seroconversion for HPV 6, 11, 16, and 18 is defined as achieving an anti-HPV cLIA level of at least 20, 16, 20 and 24 mMU/mL, respectively.
  Seroconversion rate = (number of participants with seronegative at baseline and developed seropositive at Month 7)/(number of participants with seronegative at baseline regardless relevant HPV serum status at Month 7). Measure serum anti-HPV 6, 11, 16, 18 titers at Day 1 prior to vaccination and at Month 7
Time Frame: Collect blood sample for anti-HPV 6, 11, 16, 18 titers testing at Day 1 prior to vaccination and Month 7
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Vaccine (Gardasil®) Group | Placebo Group
Number analyzed (Participants) | 302 | 298
Participants
  anti-HPV 6 | 269 | 2
  anti-HPV 11 | 279 | 2
  anti-HPV 16 | 277 | 0
  anti-HPV 18 | 287 | 3
Statistical Analysis 1: Comparison: Vaccine (Gardasil®) Group vs Placebo Group; The null hypothesis was that the seroconversion rate in the Gardasil® Group was less than 90% for each HPV type; Test type: Superiority or Other; p <= 0.05, Exact Binomial CI — The lower bound of the 95% CI for the seroconversion rate was greater than 90% for each type so the null hypothesis was rejected. The CI reported is for HPV6, the type with the smallest lower bound; Seroconversion Rate = 96.65, 95% CI [93.74 to 98.46]

3. Secondary Outcome: Serious Adverse Experiences and Systemic Adverse Experiences Occurring Within 14 Days After Each Vaccination, and Injection-site Complaints Occurring Day 1 Through Day 5 After Each Vaccination
Description: All adverse experiences were collected through 14 days following each vaccination. All participants were requested to record injection-site adverse experiences and monitor the participant's temperature daily on the Vaccination Report Card for Day 1 thereafter for 4 additional calendar days, and record all systemic adverse experiences that occur during the 14-day period after each injection.
Time Frame: For serious adverse experiences and systemic adverse experiences: 14 days follow-up after each dose of vaccination; For injection-site adverse experiences: 5 days follow-up after each dose of vaccination
Population: Safety population, defined as all participants who were vaccinated at least one dose and had safety follow-up data
Measure: Number; unit: Participants
Arm/Group | Vaccine (Gardasil®) Group | Placebo Group
Number analyzed (Participants) | 302 | 298
Participants | 153 | 131

ADVERSE EVENTS:
Arm/Group | Vaccine (Gardasil®) Group | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/302 | 1/298
Other Adverse Events (participants affected / at risk) | 260/302 | 215/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine (Gardasil®) Group (N=302) | Placebo Group (N=298)
Acute suppurative tonsillitis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1.25% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vaccine (Gardasil®) Group (N=302) | Placebo Group (N=298)
Injection site redness (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Injection site pain (Skin and subcutaneous tissue disorders) | 61 (94) | 39 (46)
Injection site induration (Skin and subcutaneous tissue disorders) | 6 (6) | 1 (1)
Injection site swelling (Skin and subcutaneous tissue disorders) | 9 (9) | 2 (3)
Injection site pruritus (Skin and subcutaneous tissue disorders) | 12 (16) | 2 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (16) | 12 (12)
Headache (Nervous system disorders) | 16 (20) | 18 (20)
Diarrhea (Gastrointestinal disorders) | 9 (11) | 10 (10)
Nausea (Gastrointestinal disorders) | 8 (9) | 12 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (12) | 10 (16)
Upper respiratory tract infection (Infections and infestations) | 18 (21) | 13 (14)
Allergic reaction (General disorders) | 8 (9) | 2 (2)
Fatigue (General disorders) | 17 (24) | 22 (25)
Fever (General disorders) | 71 (83) | 70 (85)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.